CLINICAL TRIAL: NCT06526741
Title: Alport Syndrome Foundation Alport Patient Registry
Brief Title: ASF Alport Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Alport Syndrome Foundation (Other)
Collaborators: Pulse Infoframe Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ASF-01
Record Dates: First submitted 2023-11-11; First posted 2024-07-30 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Alport Syndrome; Thin Basement Membrane Disease; Hereditary Nephritis
Keywords: Alport; COL4A3; COL4A4; COL4A5; Collagen Type-IV; Glomerulonephropathy; Glomerulosclerosis; Genetic Kidney Disease
MeSH Terms: conditions — Nephritis, Hereditary; Hematuria, Benign Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alport syndrome patients: Patients with a confirmed diagnosis of Alport syndrome by a certified genetic counselor, treating physician, or nephrologist.
  Interventions: Other: Longitudinal data collection

INTERVENTIONS:
Other: Longitudinal data collection — This is an observational ambispective non-interventional registry collecting longitudinal real-world data only. There is no intervention.

SUMMARY:
Alport Syndrome Foundation's (ASF's) Alport Patient Registry (the Registry) is open to individuals living with Alport syndrome in the United States (US) and US territories and outlying islands. The Registry welcomes participants of all ages who have a confirmed clinical diagnosis of Alport syndrome. A confirmed diagnosis could be obtained via genetic testing, biopsy, and/or from a medical professional's clinical assessment of the individual's symptoms and/or family history. Participants can have any form and stage of this disease to be eligible for inclusion in the Registry.

Patient participation in the Registry is crucial to helping attract and advance research, understanding understudied aspects of the disease, and informing clinical trials that may lead to Alport syndrome therapies and/or a cure.

The Registry is accessed through a secure, online application. Participants report their own health history in the Registry and are encouraged to update any changes, at most, every three months.

The security of each participant's information is a top priority. Any detail that could identify an individual participant is kept confidential in the Registry and such data are de-identified to protect the participant's privacy. No electronic health records or social security numbers are requested by or connected to the Registry.

A parent or legal guardian may consent to enroll a child/dren Alport patient(s) under the age of 18 years. An additional assent form is used for individuals ages 7-17. At age 18, participants will be required to re-consent as an adult if they choose to continue to participate in the Registry.

DETAILED DESCRIPTION:
ASF is an Alport syndrome patient-led 501(c)(3) non-profit based in the US. ASF regularly communicates with thousands of Alport syndrome patients, caregivers, researchers, clinicians, and industry stakeholders in the US and internationally. ASF created its Alport Patient Registry in partnership with Pulse Infoframe Inc. Together, ASF and Pulse Infoframe Inc. are committed to ensuring patients' data entered in the Registry remain secure and under the control of the patients themselves.

Alport syndrome is a genetic disease stemming from pathogenic variants in the COL4A3 gene, the COL4A4 gene (both located on the 2 chromosome), and the COL4A5 gene (located on the X chromosome). These 3 genes encode for the 3 individual collagenous strands (⍺3, ⍺4, and ⍺5 respectively) that "braid" to form the triple-helix protein collagen-typeIV⍺3,⍺4,⍺5. Collagen-typeIV⍺3,⍺4,⍺5 is an extracellular structural protein that supports and gives form and function to multiple organs and organ sub-structures in the human body including the glomeruli of the kidney, the inner ear, the eyes, skin, lungs, and blood vessels.

The primary phenotypical manifestations of Alport syndrome are:

1. Progressive glomerulonephritis leading to kidney failure. In the glomeruli of the nephrons of the kidneys, collagen-typeIV⍺3,⍺4,⍺5 is formed in specialized podocyte cells and then excreted into the extracellular matrix space between the podocytes and the endothelial (blood vessel) cells where it cross-links to form a mature glomerular basement membrane (GBM). In Alport syndrome, the GBM's structural integrity and support of podocyte viability is compromised because of the absence of healthy, functional cross-linked collagen-typeIV⍺3,⍺4,⍺5 matrix. Establishment of the cross-linked collagen-typeIV⍺3,⍺4,⍺5 matrix in the GBM starts only after birth and takes years. As such, all Alport syndrome patients are born healthy and progress to kidney failure at different rates depending on the pathogenicity of their genotype and variant. Notably, X-linked male and autosomal recessive Alport syndrome patients typically experience kidney failure in their teenage and young adult years. Also, notably, X-linked female and autosomal dominant Alport syndrome patients also suffer from kidney disease - just at a slower rate of progression - and the term "carrier" is no longer clinically accepted.
2. Often, but not always, progressive bilateral sensorineural hearing loss, particularly in the mid-to-higher frequencies.
3. Sometimes lenticonus (a bulging of the lens capsule and underlying cortex of the lenses of the eyes) and/or fleck retinopathy (yellowish-white lesions of the retinas of the eyes).
4. For patients with certain large deletion variants of the COL4A5 gene, diffuse esophageal leiomyomatoses ("benign", tumor-like growths that can cause discomfort and can interfere with swallowing).

Other phenotypical characteristics that are less understood and hypothesized include, but are not limited to, diffuse uterine leiomyomatoses, increased risk of aortic aneurysm, increased risk of preeclampsia, and the inability to recover from retinal delamination or corneal abrasions.

Because Alport syndrome stems from 3 genes that are located on both autosomal and somatic chromosomes, it exists in heterozygous, homozygous, and hemizygous forms as well as digenic and trigenic forms. Added to this complexity, pathogenic variants can present as mutations that are described as missense, nonsense, frameshift, intronic, exonic, collagenous-domain, non-collagenous-domain, or other mutations. Therefore, Alport syndrome is best characterized as a "spectrum" syndrome that encompasses tens of thousands of potential genotypical variants along with an equally diverse set of phenotypical expressions, and includes dependencies related to the patient's age, sex, treatment history, diet, and environment.

The ASF Alport Patient Registry's goals are to help understand the above described complexity of Alport syndrome by:

A) Help assessing which genetic variants influence the rate of kidney function decline.

B) Quantifying and qualifying understudied aspects of Alport syndrome.

C) Documenting medications patients are currently taking and how well they are working.

D) Supporting exploration of new therapies and potential genetic cures.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Alport syndrome by a certified genetic counselor, treating physician or nephrologist.
2. Signed informed consent/assent must be provided by the subject and/or caregiver (parent/legal guardian) including compliance with the restrictions listed in the informed consent/assent form and in the study protocol. (Separate age-appropriate assent forms are provided for ages 7-12 years and ages 13-17 years.)
3. Must reside in the USA or US territories and outlying islands. (This criterium may change at an as-yet undetermined future date.)

Exclusion Criteria:

[none]

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alport syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2048-08-23 (Estimated); Study Completion 2048-08-23 (Estimated)

PRIMARY OUTCOMES:
Total number of enrolled participants | 5 years
  Reach 750 enrolled participants

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A Weinstock, PhD, Principal Investigator — Alport Syndrome Foundation
Locations (1):
- On-line only: https://asfalportpatientregistry.healthie.net, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Agreement between the ASF and Pulse Infoframe based on Pulse Infoframe's models for other rare disease registries they have supported.

REFERENCES:
- See also: ASF Alport Patient Registry new registration link — https://asfalportpatientregistry.healthie.net/register
- See also: ASF Alport Patient Registry returning participant/legal guardian login — https://asfalportpatientregistry.healthie.net/login
- See also: Alport Syndrome Foundation (sponsor) — https://alportsyndrome.org
- See also: Pulse Infoframe Inc. (partner & host) — https://www.pulseinfoframe.com
- See also: North Star Review Board (independent review board) — https://learningirb.org

DOCUMENTS (2):
  • Study Protocol (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT06526741/Prot_000.pdf
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT06526741/ICF_001.pdf